CLINICAL TRIAL: NCT02188589
Title: Evaluation of an Absorbable Implant for the Treatment of Nasal Valve Collapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spirox, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPI-NVC-13001
Record Dates: First submitted 2014-07-04; First posted 2014-07-11 (Estimated); Results first posted 2016-10-10 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2018-11

CONDITIONS: Nasal Valve Collapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nasal implant group (Experimental): Bilateral or unilateral INEX nasal implants
  Interventions: Device: INEX nasal implant

INTERVENTIONS:
Device: INEX nasal implant — Treatment group may receive unilateral or bilateral INEX nasal implants (maximum of 4, 2 per side)

SUMMARY:
To evaluate the safety and feasibility of the INEX Nasal Implant in subjects with moderate to severe nasal valve collapse.

DETAILED DESCRIPTION:
This study is a multicenter, nonrandomized, prospective exploratory study of the INEX Nasal Implant. The purpose of this study is to evaluate the safety and feasibility of the INEX Nasal Implant in subjects with moderate to severe nasal valve collapse.

ELIGIBILITY:
Eligible participants are:

1. Adult patients seeking treatment for nasal obstruction on one or both sides of the nose who are willing to undergo an office-based or intraoperative nasal implant procedure in lieu of alternative treatments (ie, surgical repair or use of an external dilator).
2. Nasal valve collapse (NVC) must be a primary or significant contributor to the subject's nasal obstruction based on clinical presentation, physical examination and nasal endoscopy.
3. Baseline Nasal Obstruction Symptom Evaluation (NOSE) score must be ≥55.

Participants are excluded for the following:

1. Surgical or non-surgical treatment of the nasal valve or rhinoplasty within 12 months before enrollment.
2. Septoplasty, inferior turbinate reduction, or other surgical nasal procedures within 6 months before enrollment.
3. Recurrent nasal infections.
4. Use of intranasal steroids within 2 weeks preimplant and 2 weeks post implantation.
5. Presence of a permanent implant, dilator, or uses an external device in the nasal area.
6. Cancerous or precancerous lesions and/or radiation exposure in the treatment area or chemotherapy within 24 months of the study.
7. Significant bleeding disorders.
8. Significant systemic diseases.
9. Currently using nasal oxygen or continuous positive airway pressure (CPAP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Berghaus, MD, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Klinik und Poliklinik für Hals-Nasen-Ohren-Heilkunde am Klinikum der LMU, Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stewart MG, Witsell DL, Smith TL, Weaver EM, Yueh B, Hannley MT. Development and validation of the Nasal Obstruction Symptom Evaluation (NOSE) scale. Otolaryngol Head Neck Surg. 2004 Feb;130(2):157-63. doi: 10.1016/j.otohns.2003.09.016. PMID 14990910
- [Result] San Nicolo M, Stelter K, Sadick H, Bas M, Berghaus A. Absorbable Implant to Treat Nasal Valve Collapse. Facial Plast Surg. 2017 Apr;33(2):233-240. doi: 10.1055/s-0037-1598655. Epub 2017 Apr 7. PMID 28388804
- [Result] San Nicolo M, Stelter K, Sadick H, Bas M, Berghaus A. A 2-Year Follow-up Study of an Absorbable Implant to Treat Nasal Valve Collapse. Facial Plast Surg. 2018 Oct;34(5):545-550. doi: 10.1055/s-0038-1672213. Epub 2018 Sep 18. PMID 30227454

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Nasal implant: Treatment group may receive unilateral or bilateral nasal implants (maximum of 4, 2 per side)
Period: Overall Study
Arm/Group | Treatment Group
Started | 30
6 Months | 30
12 Months (Final follow-up under initial protocol.) | 30
24 Months (Extended follow-up protocol, participants signed additional consent for follow-up beyond 12 months.) | 25
Completed | 25
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Implant-related Adverse Events
Description: Implant-related adverse events (such as implant retrievals, procedure-related hematoma/inflammation)
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 30
participants | 5

2. Secondary Outcome: Breathing Capacity (NOSE Scores)
Description: Nasal breathing capacity was assessed using the validated Nasal Obstruction Symptom Evaluation (NOSE) questionnaire. The NOSE score uses a 0-100 point scale to capture severity of nasal symptoms (congestion, obstruction, trouble breathing, sleeping, and exercise), with higher scores indicating more severe symptoms than lower scores. NOSE severity classes are defined as Mild (5-25), Moderate (30-50), Severe (55-75), and Extreme (80-100).
Time Frame: At baseline and at 6, 12, and 24 months post implant
Population: All 30 participants completed follow-up through 12 months. Five participants discontinued after the 12-month visit and before the 24-month visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 30
scores on a scale
  Baseline | 76.7 (14.8)
  6 Months | 33.3 (29.7)
  12 Months | 35.2 (29.2)
  24 Months: number analyzed (Participants) | 25
  24 Months | 32.0 (29.3)
Statistical Analysis 1: Comparison: Treatment Group; Test type: Equivalence — The difference between the mean baseline and mean follow-up NOSE scores was evaluated by paired t-test with significance indicated by p<0.05; p < 0.001, t-test, 2 sided

3. Secondary Outcome: NOSE Responder Rate
Description: Percent of participants meeting responder criteria. Responders are defined as participants with a reduction from baseline in 1 or more Nasal Obstruction Symptom Evaluation Score (NOSE) severity class or a 20% reduction in the NOSE score.
Time Frame: At 6, 12, and 24 months post implant
Population: as for outcome 2
Measure: Number; unit: percentage of responders
Groups:
- Nasal Implant Group: Treatment group may receive unilateral or bilateral INEX nasal implants (maximum of 4, 2 per side)
Arm/Group | Nasal Implant Group
Number analyzed (Participants) | 30
percentage of responders
  6 Months | 80.0
  12 Months | 76.7
  24 Months: number analyzed (Participants) | 25
  24 Months | 80.0

ADVERSE EVENTS:
Time Frame: Through 24 months post implant
Description: Device extrusions/retrievals were counted as serious implant-related adverse events. Otherwise, the standard definition applies.
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 5/30
Other Adverse Events (participants affected / at risk) | 10/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=30)
Nonsurgical implant retrieval (Investigations) | 3 (3) — 3/56 total implants placed were retrieved post implantation. Implant retrieval did not require surgical intervention and did not result in any adverse clinical sequelae.
Hernia Repair Procedure (Surgical and medical procedures) | 1 (1) — Hernia repair procedure occurred during the follow-up period and was not related to the investigational device or the nasal implant procedure.
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Bronchitis occurred during the follow-up period and was not related to the investigational device or the nasal implant procedure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=30)
Hematoma (Skin and subcutaneous tissue disorders) | 1 (1) — A non-serious device-related hematoma was observed.
Inflammation (Skin and subcutaneous tissue disorders) | 1 (1) — A non-serious device-related observation of inflammation was reported.
Rhinitis (General disorders) | 3 (3) — Includes reports of rhinitis and "common cold", non-serious and not device-related
Rhinorrhea (General disorders) | 2 (2) — Non-serious and not device-related
Acute hypertension (Vascular disorders) | 1 (1) — Non-serious and not device-related
Injury by fallen tree (Social circumstances) | 1 (1) — Non-serious and not device-related
Vertigo (General disorders) | 1 (1) — Non-serious and not device-related
Headache (General disorders) | 1 (1) — Non serious and not device-related
Normal Bleeding Epistaxis (Blood and lymphatic system disorders) | 1 (1) — Normal bleeding epistaxis occurred during the follow-up period and was not related to the investigational device or the nasal implant procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No